CLINICAL TRIAL: NCT02815826
Title: 16 Weeks of Progressive Barefoot Running Training Changes Impact Force and Muscle Activation in Habitual Shod Runners
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ana Paula da Silva Azevedo, Principal Investigator, University of Sao Paulo
Other Study IDs: EEFEUSP_LBiomec-1
Record Dates: First submitted 2016-06-22; First posted 2016-06-28 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Barefoot Running

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Barefoot training: 16 weeks of progressive barefoot running training
  Interventions: Other: Barefoot training; Other: Shod training

INTERVENTIONS:
Other: Barefoot training — During 16 weeks, habitual shod runners kept their normal running training routine (wearing shoes), while they were introduced progressively to BF condition. Three training sessions were performed per week. Barefoot training started with 5% and ended with 20% of their WTV being performed without shoes. Soft surfaces (i.e. sand and grass) were adopted in the beginning of training (week 1 to 8). From week 9 to 16, participants mixed soft with harder surfaces, as treadmill and asphalt, to accomplish the training.
Other: Shod training — Running training planned individually to each runner, according to their physical fitness, and performed with shoes.

SUMMARY:
The purpose of this study was to evaluate the influence of 16 weeks of progressive barefoot running training on impact force and muscle activation in habitual shod runners. Habitual shod runners were tested barefoot (BF) and shod (SH), before and after 16 weeks of progressive barefoot running training. Tests consisted of running on instrumented treadmill at 9 km/h, for 10 minutes in each experimental condition. Nine data acquisitions (10 s) of vertical ground reaction force (VGRF) and electromyographic (EMG) signal were conducted in each experimental condition, for each test.

DETAILED DESCRIPTION:
Short-term effects of barefoot and simulated barefoot running have been widely discussed in recent years. Consequences of adopting barefoot running for a long period, e.g. as training strategy, still remain unknown. The present study evaluated the influence of 16 weeks of progressive barefoot running training on impact force and muscle activation in habitual shod runners. Habitual shod runners were tested barefoot (BF) and shod (SH), before and after 16 weeks of progressive barefoot running training. During the 16 weeks of training, participants kept their normal running training routine (wearing shoes), while they were introduced progressively to BF condition. Three training sessions were performed per week. Barefoot training started with 5% and ended with 20% of their weekly training volume (WTV) being performed without shoes. Soft surfaces (i.e. sand and grass) were adopted in the beginning of training (week 1 to 8). From week 9 to 16, participants mixed soft with harder surfaces, as treadmill and asphalt, to accomplish the training. Training sessions were prepared by professionals, researches and participants together. All training sessions were supervised by the researchers. Tests consisted of running on instrumented treadmill at 9 km/h, for 10 minutes in each experimental condition. Each session test started with participants performing a maximum voluntary isometric contraction (MVIC) test for each muscle of interest. The MVIC protocol consisted of 4 movement trials for each muscle: 2 submaximal trials of 10 seconds; 1 maximal trial of 5 seconds; and 1 maximal trial of 10 seconds. Then, a 5-minute period of warm-up at self-selected speed was performed on a treadmill. After that, participants ran (at 9km/h) during 10 minutes on an instrumented treadmill in both barefoot and shod conditions. Participants had a 2-minute interval between each trial while experimental condition was changed. The VGRF of both legs and EMG signal of tibialis anterior (TA), gastrocnemius lateralis (GL), long head of biceps femoris (BCF), rectus femoris (RF) and vastus lateralis (VL) of the right leg of each volunteer were obtained. These muscles were chosen due to their importance and contribution to running. For shod trial, runners wore their own habitual running shoes. All shoes were in good conditions of use and had similar characteristics of construction.

ELIGIBILITY:
Inclusion Criteria:

* to have a minimum of 6 months of regular running training;
* to have a minimum of 6 months of experience in running on treadmills;
* do not have suffered any orthopedic injury in the last 12 months.

Exclusion Criteria:

* to have experience in minimalist/barefoot running;
* to be habitual forefoot striker;
* to complete less than 80% of training;
* to suffer any injury during training.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Habitual shod runners (recreational runners without experience in barefoot and/or minimatist running)
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2012-09; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Parameters of the vertical component of Ground Reaction Force (VGRF) related to impact force | 4 months
  Biomechanical parameters related to impact forces, as magnitude of VGRF's first peak, time to reach first peak of VGRF and implulse from the first 50 ms, will be measured.
Electromyographic (EMG) parameters related to muscle activation intensity | 4 months
  EMG signal will be measeured and the RMS, a parameter that reflects muscle activation intensity, will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Ana Paula da Silva Azevedo, São Paulo, São Paulo, Brazil